CLINICAL TRIAL: NCT02393196
Title: Colloid Preload Versus Colloid Coload in Preventing Spinal Anesthesia-Induced Hypotension During Cesarean Section Deliveries: A Prospective, Randomized, Double-Blind Comparative Study
Brief Title: Colloid Preload Versus Colloid Coload During Cesarean Deliveries
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sifa University (Other)
Responsible Party: Principal Investigator, Aysun Afife Kar, Assistant Professor, Sifa University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SifaU
Record Dates: First submitted 2015-03-01; First posted 2015-03-19 (Estimated); Last update posted 2015-11-17 (Estimated); Status verified 2015-11

CONDITIONS: Anesthesia; Adverse Effect, Spinal and Epidural; Hypotension
Keywords: colloid preloading; colloid coloading
MeSH Terms: conditions — Hypotension | interventions — Hydroxyethyl Starch Derivatives; HES 130-0.4

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group Preloading (Group P) (Active Comparator): Group Preloading (Group P): 500 mL hydroxyethyl starch (6% HES 130/0.4) (Voluven®; Fresenius Kabi, Bad Homburg, Germany) will be infused via a pressure infusion system at a maximum speed as possible before spinal anesthesia.
  Interventions: Drug: hydroxyethyl starch (% 6 HES 130/0.4) (Voluven®)
- Group Coloading (Group C) (Active Comparator): Group Coloading (Group C): After the patients have been monitored, spinal anesthesia will be performed. Recognizing the cerebrospinal fluid, 500 mL hydroxyethyl starch (%6 HES 130/0.4) (Voluven®; Fresenius Kabi, Bad Homburg, Germany) will be infused via a pressure infusion system at a maximum speed as possible.
  Interventions: Drug: hydroxyethyl starch (%6 HES 130/0.4) (Voluven®)

INTERVENTIONS:
Drug: hydroxyethyl starch (% 6 HES 130/0.4) (Voluven®) — Before spinal anesthesia
  Other Names: (Voluven®; Fresenius Kabi, Bad Homburg, Germany)
  Arms: Group Preloading (Group P)
Drug: hydroxyethyl starch (%6 HES 130/0.4) (Voluven®) — Just after spinal anesthesia
  Other Names: (Voluven®; Fresenius Kabi, Bad Homburg, Germany)
  Arms: Group Coloading (Group C)

SUMMARY:
The investigators aimed to compare the methods colloid preloading and colloid coloading in terms of the incidence of maternal hypotension and impacts on neonatal outcomes. The second aim while planning the present study is to identify the method of the lowest adverse event for mother and infant and the simplest approach for the clinician.

DETAILED DESCRIPTION:
Spinal anesthesia (SA) is currently the most preferred method of anesthesia in elective cesarean deliveries. However, SA causes maternal hypotension by decreasing systemic vascular resistance over sympathetic blockade. Maternal hypotension can lead to serious adverse events both in mother and in fetus: fetal hypoxia and acidosis occur due to decreased uterine blood flow, whereas the mother may experience vertigo, nausea, vomiting, alteration in consciousness, cardiovascular collapse and arrest. Today, various strategies have been suggested for the prevention of maternal hypotension. Of these strategies, the most critical ones are fluid load before spinal anesthesia (preloading) or rapid fluid load just after spinal anesthesia (coloading) and the use of vasopressor agent. The fluids used for this purpose include crystalloids and colloids. Comparative studies performed with colloid preloading, colloid coloading and crystalloid coloading indicated that the incidence of hypotension decreased similarly with no significant difference determined between the methods of fluid loading. Researchers defended necessity of using vasopressor agent together with fluid loading methods. In daily routine; however, the investigators observe that the incidence of hypotension is lower in the patients that undergo colloid preloading as compared to the patients that undergo colloid coloading or crystalloid coloading. The investigators therefore aimed to compare the methods colloid preloading and colloid coloading in terms of the incidence of maternal hypotension and impacts on neonatal outcomes. In the present study, the investigators aimed to use 6% HES 130/0.4 (Voluven ®), which is the newer generation colloid solution. The other aim while planning the present study is to identify the method of the lowest adverse event for mother and infant and the simplest approach for the clinician.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Singleton pregnancy
* Gestational age ≥ 37 weeks
* Height ≥ 150 cm and ≤ 180 cm
* Weight > 50 kg and < 100 kg

Exclusion Criteria:

* Gestational age > 37 weeks
* Multiple pregnancies
* Fetal distress
* Preeclampsia
* Cardiovascular disease and diabetes
* Hematological problems
* Local infection at intervention site
* Abnormal coagulation tests
* Anticoagulant use
* Starch allergy
* Height < 150 cm and > 180 cm
* Weight < 50 kg and > 100 kg

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2015-03; Primary Completion 2016-01 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Maternal hypotension. | Time between induction of spinal anesthesia until delivery (umbilical cord clamping). Participants will be followed for the duration of hospital stay, an expected average of two days.
  Maternal hypotension will be defined as at least a single administration of ephedrine within the period from induction of SA to the delivery (umbilical cord clamping). After spinal anesthesia, SAP will be measured and recorded at every minute until birth and every three minutes thereafter.
Incidence of severe hypotension. | Time between induction of spinal anesthesia until delivery (umbilical cord clamping). Participants will be followed for the duration of hospital stay, an expected average of two days.
  Incidence of severe hypotension (SAP < 70% of the baseline value or SAP < 80 mmHg) will be recorded.
Cumulative duration of hypotension. | Time between induction of spinal anesthesia until delivery (umbilical cord clamping). Participants will be followed for the duration of hospital stay, an expected average of two days.
  Cumulative duration of hypotension will be recorded from induction of spinal anesthesia until delivery (umbilical cord clamping).
Heart rate. | Time between induction of spinal anesthesia until delivery (umbilical cord clamping). Participants will be followed for the duration of hospital stay, an expected average of two days.
  Minimum and maximum heart rate, bradycardia, atropine usage will be recorded.

SECONDARY OUTCOMES:
Neonatal effects. | Time just after delivery (umbilical cord clamping). Participants will be followed for the duration of hospital stay, an expected average of two days.
  Arterial and venous blood gas analyses will be performed from the umbilical cord after the cord clamped.
Ephedrine treatment. | Time between induction of spinal anesthesia until delivery (umbilical cord clamping). Participants will be followed for the duration of hospital stay, an expected average of two days.
  If SAB < 100 mmHg; patients will be treated by 5 mg IV bolus ephedrine, if SAB < 90 mmHg; patients will be treated by 10 mg IV bolus ephedrine.
Nausea and/or vomiting. | Time between induction of spinal anesthesia until delivery (umbilical cord clamping). Participants will be followed for the duration of hospital stay, an expected average of two days.
  Incidence of nausea and/or vomiting, incidence of prepartum nausea and/or vomiting will be recorded.

OTHER OUTCOMES:
Preoperative fasting period. | Time before spinal anesthesia. Participants will be followed for the duration of hospital stay, an expected average of two days.
  preoperative fasting period will be recorded.
Preoperative hemoglobin concentration (g/dL). | Time before spinal anesthesia. Participants will be followed for the duration of hospital stay, an expected average of two days.
  Before spinal anesthesia. Participants will be followed for the duration of hospital stay, an expected average of two days.
Durations of anesthesia and surgery. | Time between induction of spinal anesthesia until end of the anesthesia. Participants will be followed for the duration of hospital stay, an expected average of two days.
  Time period from induction of spinal anesthesia to skin incision (min), time period from induction of spinal anesthesia to delivery (min), time period from uterine incision to birth (sec), duration of anesthesia (min), and duration of surgery (min) will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Aysun Afife Kar, MD, Principal Investigator — Şifa Üniversitesi, Basmane Hastanesi, İzmir, Turkey
Locations (1):
- Şifa Üniversitesi, Basmane Hastanesi, Izmir, Turkey (Türkiye)